CLINICAL TRIAL: NCT01521000
Title: The Use of Bioimpedance to Determine Pre-Clinical Lymphedema in the Post-Operative Breast Cancer Patient
Acronym: L-Dex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Main Line Health (Other)
Collaborators: Sharpe-Strumia Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F/N-R10-2932B
Record Dates: First submitted 2011-02-09; First posted 2012-01-30 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Lymphedema; Sentinel Node Biopsy; Axillary Dissection
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation (No Intervention): Observation arm will continue to be followed with serial L-Dex and water volume displacement methods.
  Interventions: Device: Garment Sleeve
- Intervention-garment sleeve (Other): If the L-Dex is outside the normal range, or has increased 10 units from baseline, the patient will then be randomized to wear a compression sleeve (20 to 30 mm of Hg) daily for 4 weeks or observation (no sleeve). After 4 weeks, L-Dex measurements and water volume displacement will be reassessed in the treatment group.
  Interventions: Device: Garment Sleeve

INTERVENTIONS:
Device: Garment Sleeve — compression sleeve (20 to 30 mm of Hg)

SUMMARY:
Primary Objective: To determine whether early intervention (with garment sleeve and gauntlet) in patients with pre-clinical lymphedema can halt the progression of lymphedema.

Secondary Objectives:To evaluate whether bioimpedance is an accurate, reliable method to measure pre-clinical and clinical lymphedema.

Tertiary Objective: To determine whether bioimpedance analysis is better than the gold standard of volume displacement to measure lymphedema.

The successful completion of this study will address whether bioimpedance analysis is a reliable, accurate method to measure pre-clinical and clinical lymphedema. In addition, we intend to evaluate whether bioimpedance analysis is better than the gold standard of volume displacement for measuring lymphedema. And most importantly, we will evaluate whether a short trial of compression garments in women identified to have pre-clinical lymphedema can actually halt the progression of disease. Bryn Mawr Hospital would propose to publish the research and findings of this study, which may have future bearing on the post-operative therapeutic management of subjects with pre-clinical lymphedema following axillary surgery.

Study Design:Randomized, Pilot Study

DETAILED DESCRIPTION:
Primary Objective: To determine whether early intervention (with garment sleeve and gauntlet) in patients with pre-clinical lymphedema can halt the progression of lymphedema.

Secondary Objectives:To evaluate whether bioimpedance is an accurate, reliable method to measure pre-clinical and clinical lymphedema.

Tertiary Objective: To determine whether bioimpedance analysis is better than the gold standard of volume displacement to measure lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* are female
* have operable, early stage breast cancer stage 0 - IIIA
* undergo axillary evaluation with either sentinel lymph node biopsy or axillary lymph node dissection
* are aged > 18 years of age at the date of enrollment
* are willing to sign an informed consent form

Exclusion Criteria:

* are male
* have had a bilateral axillary surgery
* do not undergo axillary evaluation
* are a minor
* cannot consider the issues involved in making an informed and autonomous decision.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To determine whether early intervention in patients with pre-clinical lymphedema can halt the progression of lymphedema. | 2 years
  Evaluate whether a short trial of compression garments in women identified to have pre-clinical lymphedema can actually halt the progression of disease.

SECONDARY OUTCOMES:
200 women will have bioimpedance and volume displacement measurements to evaluate whether bioimpedance is an accurate, reliable method to measure pre-clinical and clinical lymphedema as compared to standard (volume displacement) | 2 years
  Evaluate whether bioimpedance analysis is better than the gold standard of volume displacement for measuring lymphedema.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea V Barrio, MD, Principal Investigator — Bryn Mawr Hospital
Locations (1):
- Comprehensive Breast Center at Bryn Mawr Hospital, Bryn Mawr, Pennsylvania, United States